CLINICAL TRIAL: NCT04013542
Title: A Pilot Trial of Ipilimumab-Nivolumab in Local-Regionally Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: Ipilimumab and Nivolumab in Combination With Radiation Therapy in Treating Patients With Stage 2-3 Non-small Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0836; NCI-2019-03205 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0836 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-08; First posted 2019-07-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: ALK Gene Rearrangement; EGFR Gene Mutation; Locally Advanced Lung Non-Small Cell Carcinoma; Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ipilimumab, radiation therapy) (Experimental): CONCURRENT THERAPY: Patients receive nivolumab IV over 30 minutes on day 1 and ipilimumab IV over 30 minutes on day 1. Treatment with nivolumab repeats every 21 days for up to 8 cycles, and treatment with ipilimumab repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 1 day of starting nivolumab and ipilimumab, patients also undergo radiation therapy 5 days a week (Monday-Friday) over 6-7 weeks in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase I trial studies the side effects of ipilimumab and nivolumab in combination with radiation therapy, and to see how well they work in treating patients with stage II-III non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy rays to kill tumor cells and shrink tumors. Ipilimumab and nivolumab may also help radiation therapy work better by making tumor cells more sensitive to the radiation therapy. Giving ipilimumab and nivolumab in combination with radiation therapy may work better in treating patients with stage II-III non-small cell lung cancer compared to standard chemotherapy in combination with radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine safety and feasibility of ipilimumab-nivolumab (Bristol-Meyers-Squibb, Opdivo), a cytotoxic T-lymphocyte-associated protein 4 (CTLA4) and programmed death 1 (PD-1) inhibitor in the treatment of local-regionally advanced non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate the clinical outcomes of treatment with ipilimumab-nivolumab concurrent with radiation therapy in patients with local-regionally advanced NSCLC.

II. To observe and record anti-tumor activity. III. To identify potential predictive and prognostic biomarkers for early recurrence using circulating cell-free deoxyribonucleic acid (DNA) (cfDNA).

IV. To identify potential predictive and prognostic biomarkers for early recurrence using tumor tissue PD-L1 immunohistochemistry (IHC).

V. To identify potential predictive and prognostic biomarkers for early recurrence using tumor tissue tumor mutational burden (TMB).

VI. To identify potential resistance mechanisms using immune biomarker and genetic analysis in post-progression biopsies.

EXPLORATORY OBJECTIVES:

I. Tumor tissue/blood biomarkers will be assessed for tumor mutation burden (TMB) and PD-L1 immunohistochemistry.

II. Patient microbiomes will be evaluated with stool specimen collection kits.

OUTLINE:

CONCURRENT THERAPY: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and ipilimumab IV over 30 minutes on day 1. Treatment with nivolumab repeats every 21 days for up to 8 cycles, and treatment with ipilimumab repeats every 42 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Within 1 day of starting nivolumab and ipilimumab, patients also undergo radiation therapy 5 days a week (Monday-Friday) over 6-7 weeks in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed NSCLC (any histology)
* Patients must have stage II or III local-regionally advanced NSCLC that is deemed to be best treated by systemic and concurrent radiotherapy. Eligible patients with stage II disease must be unresectable or refuse surgical resection
* No prior therapy for the current stage II or stage III NSCLC disease
* ECOG (Eastern Cooperative Oncology Group) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.5 x institutional ULN
* Glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* No prior history of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
* No prior history of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computerized tomography (CT) scan
* No active pregnancy. The effects of ipilimumab-nivolumab on the developing human fetus are unknown. For this reason and because radiation and possibly immunotherapies used in this trial are known or possibly known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 months after completion of ipilimumab-nivolumab administration
* Ability to understand and the willingness to sign a written informed consent document
* Patients with known epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) rearrangement are eligible

Exclusion Criteria:

* Prior systemic therapy for the current active local-regionally advanced NSCLC
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because nivolumab is an immunotherapy agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, breastfeeding should be discontinued if the mother is treated with nivolumab. These potential risks may also apply to radiation therapy used in this study
* Known human immunodeficiency virus (HIV) positivity
* Active chronic treatment (that is still required) with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents)
* Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Active untreated hepatitis. Patients with known past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA (ribonucleic acid). Hepatitis B virus (HBV) and HCV viral loads must also be undetectable
* Known active untreated tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks before treatment start or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to treatment start or at any time during the study
* Malignancies within 3 years prior to treatment start, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated stage I-II cancers, carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., CLL [chronic lymphocytic leukemia] Rai stage 0, prostate cancer with Gleason score =< 6, and prostate-specific antigen [PSA] =< 10 mg/mL, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Safety and tolerability will be assessed by the incidence and severity of adverse events as determined by Common Terminology Criteria for Adverse Events version 5 and by physical examination findings, clinical laboratory tests, and vital signs, assessments.

SECONDARY OUTCOMES:
Anti-tumor activity | Up to 2 years
  The anti-tumor activity of study treatment will be assessed by the site investigators according to the Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1).
Progression-free survival (PFS) | Up to 2 years
  Will be evaluated using the method of Kaplan-Meier. Confidence intervals around the median will be calculated using the Brookmeyer-Crowley method.
Overall survival (OS) | Up to 2 years
  Will be evaluated using the method of Kaplan-Meier. Confidence intervals around the median will be calculated using the Brookmeyer-Crowley method.
Time to local treatment failure | Up to 2 years
  Will be evaluated using the method of Kaplan-Meier. Confidence intervals around the median will be calculated using the Brookmeyer-Crowley method.
Time to distant treatment failure | Up to 2 years
  Will be evaluated using the method of Kaplan-Meier. Confidence intervals around the median will be calculated using the Brookmeyer-Crowley method.
Overall response rate | Up to 2 years
Duration of response | Up to 2 years

OTHER OUTCOMES:
Tumor tissue/blood biomarkers | Up to 2 years
  Will be assessed for tumor mutational burden and PD-L1 immunohistochemistry and will be correlated to clinical outcomes of response, PFS, and OS. Biomarker effects will be summarized using descriptive statistics and associations with clinical efficacy and/or safety outcomes may be explored.
Microbiome evaluation | Up to 2 years
  The microbiome flora will be correlated to clinical outcomes of response, PFS, and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Tsao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT04013542/ICF_000.pdf